CLINICAL TRIAL: NCT01239017
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group, Single Dose Study of the Safety and Efficacy of Subcutaneously Administered REGN475 in Patients With Osteoarthritis of the Knee
Brief Title: A Study of the Safety and Efficacy of Subcutaneously Administered REGN475 in Patients With Osteoarthritis of the Knee
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Paul Tiseo, PhD - Medical Director, Regeneron Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R475-PN-1004
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose 1 (Experimental): SC REGN475 Dose 1 and IV Placebo
  Interventions: Biological: REGN475
- Dose 2 (Experimental): SC REGN475 Dose 2 and IV Placebo
  Interventions: Biological: REGN475
- Dose 3 (Experimental): SC REGN475 Dose 3 and IV Placebo
  Interventions: Biological: REGN475
- Dose 4 (Experimental): SC Placebo and IV REGN475 Dose 4
  Interventions: Biological: REGN475
- Dose 5 (Placebo Comparator): SC Placebo and IV Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: REGN475
  Arms: Dose 1; Dose 2; Dose 3; Dose 4
Other: Placebo
  Arms: Dose 5

SUMMARY:
This is a double-blind, prospective, randomized study in which patients will be randomized to 1 of 5 treatment arms (4 active and 1 placebo).

Each patient will receive one SC injection of REGN475 or placebo and 1 IV infusion of either REGN475 or placebo, on day 1 (baseline) In order to preserve the blind, patients receiving REGN475 SC will also receive placebo IV, and patients receiving REGN475 IV will also receive placebo SC.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of OA of the knee according to American College of Rheumatology (ACR) criteria, and experiencing moderate to severe pain in the index knee for at least 3 months prior to the screening visit.
2. Kellgren-Lawrence grade 2-3 radiographic severity of the index knee at or within 6 months prior to Screening.

Exclusion Criteria:

1. Significant concomitant illness including, but not limited to, cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease that would adversely affect the patient's participation in the study.
2. Patients with joint replacement in the affected knee.
3. Intra-articular injection of corticosteroids or hyaluronic acid in the affected knee within the 3 months prior to the screening visit.
4. Women who are pregnant or breast-feeding.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events (TEAEs) in patients treated with REGN475 or placebo. | 16 weeks

SECONDARY OUTCOMES:
Time-integrated change from baseline in walking knee pain using the Numeric Rating Scale (NRS). | 8 weeks
Change from baseline in walking knee pain using the Numeric Rating Scale (NRS). | 8 weeks
Time-integrated change from baseline in The Western Ontario and McMaster Osteoarthritis Index (WOMAC) | 8 weeks
Change from baseline in The Western Ontario and McMaster Osteoarthritis Index (WOMAC) | 8 weeks
Patient assessment of response to treatment over time using the Patient Global Impression of Change. | 16 weeks
Change from baseline in patient-rated QOL using the Short-Form 12-Item Questionnaire (SF-12). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Tiseo, PhD, Study Director — Regeneron Pharmaceuticals